CLINICAL TRIAL: NCT05359198
Title: Patient Reported Outcome Study on Long Term LoFric Users
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: LOF-0027
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Urinary Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
A prospective, observational cohort study evaluating Patient Reported Outcome in subjects with a long term experience from intermittent catheterization using the LoFric catheter. Prescription and use of LoFric catheters fall within current practice and is not dictated within this Non-Interventional Study.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent.
2. Female or male aged 18 years or older at time of signing informed consent.
3. Use of LoFric catheters for urethral intermittent catheterization for ≥ 6 years and currently using LoFric.
4. Able to read and write.
5. By investigator judged as able to comprehend and answer study questionnaires.

Exclusion Criteria:

1. Use of other catheter brand(s) than LoFric for > 8 weeks in total during the past 12 months.
2. Simultaneous participation in any interfering clinical study as judged by the investigator.
3. Involvement in the planning and/or conduct of the NIS (applies to both Wellspect HealthCare staff and staff at the study site).
4. Previous enrolment in the present NIS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women, aged 18 years or above, practicing urethral intermittent catheterization. The patients should have used LoFric catheters ≥ 6 years for the purpose of urethral intermittent catheterization.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-10-08 (Estimated)

PRIMARY OUTCOMES:
Document urological complications | 5 years
  Number of UTIs last 12 months
Document urological complications | 5 years
  Hospitalization due to UTI last 12 months
Document urological complications | 5 years
  Urethral stricture last 12 months
Document urological complications | 5 years
  Reflux last 12 months
Document urological complications | 5 years
  Urosepsis last 12 months
Document urological complications | 5 years
  Prostatitis last 12 months
Document urological complications | 5 years
  Epididymitis last 12 months
Document urological complications | 5 years
  Bladder stone(s) last 12 months
Document urological complications | 5 years
  Incontinence
Document urological complications | 5 years
  Other urological complications last 12 months
Quality of Life Data | 5 years
  EQ-5D variables QoL data will be collected at each measuring point using the validated instrument EQ-5D-3L (EQ-5D). The EQ-5D, consisting of a questionnaire and a visual analogue scale (VAS), is a standardized health-related quality of life questionnaire developed by the EuroQoL Group in order to provide a simple, generic measure of health for clinical and economic appraisal. The VAS is a self-rated health status scale and records the subject's perception of his/her own current overall health and can be used to monitor changes over time. The questionnaire is a self-reported description of the subject's current health in 5 dimensions; mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The subject is asked to grade their own current level of function in each dimension on a three-graded scale (i.e. no problems, some problems or severe problems) and the combination of these creates a unique health state.
Patient perception of therapy | 5 years
  PRO variables Four questions regarding perception of subject's intermittent catheter therapy. Response on a 4 graded scale; Strongly agree, agree, disagree, strongly disagree.
  Changes will be followed during study period.
Patient perception of LoFric | 5 years
  PRO variables Eight questions regarding perception of subject's catheter. Response on a 4 graded scale; Strongly agree, agree, disagree, strongly disagree.
  Changes will be followed during study period.
Compliance/non-compliance to LoFric | 5 years
  PRO variables Type of catheter used collected during study period